CLINICAL TRIAL: NCT07337239
Title: Assessment of the Effect of Hypoglossal Nerve Stimulation Therapy on Upper Airway Collapsibility During Drug-induced Sleep Endoscopy
Acronym: HNS-CoDSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8169
Record Dates: First submitted 2025-11-25; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; DISE; Endotyping; Collapsibility
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Patients who undergo hypoglossal nerve stimulation therapy will be recruited at the one year follow-up appointment at the department of ENT. As part of the standard clinical pathway, these patients will have a PSG and DISE planned one year after HNS-therapy intiation. Participants of this study will be invited to to have their one year follow-up DISE extended with additional measurements to assess the effect of HNS therapy on upper airway collapsibility.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DISE extended with additional measurements (Experimental): Patients who undergo hypoglossal nerve stimulation therapy will be recruited at the one year follow-up appointment at the department of ENT. As part of the standard clinical pathway, these patients will have a PSG and DISE planned one year after HNS-therapy intiation. Participants of this study will be invited to to have their one year follow-up DISE extended with additional measurements to assess the effect of HNS therapy on upper airway collapsibility.
  Interventions: Procedure: Additional measurements during clinical standard follow-up drug-induced sleep endoscopy (DISE)

INTERVENTIONS:
Procedure: Additional measurements during clinical standard follow-up drug-induced sleep endoscopy (DISE) — During standard DISE, type I polysomnography (Alice LDx 6, Philips Respironics) expanded with measurements of Pcrit (Pcrit3000 device, Philips Respironics) and airflow (Pneumotachometer, Hans-Rudolph, USA) will be performed.

SUMMARY:
This clinical trial will evaluate the effect of treatment with hypoglossal nerve stimulation on the underlying mechanisms of obstructive sleep apnea. Several disease mechanism parameters are known to be associated with obstructive sleep apnea. However, currently, only the location of upper airway collapse is routinely examined in clinical practice using sleep endoscopy. Among other parameters, airway collapsibility is a widely studied mechanism. This parameter indicates how easily a patient's upper airway tends to collapse and can be assessed with additional measurements during sleep endoscopy.

The aim of this trial is to investigate the effect of hypoglossal nerve stimulation on collapsibility during sleep endoscopy. This information will provide a better understanding of the physiological mechanisms of hypoglossal nerve stimulation. In the long term, the investigators hope this knowledge will allow for more personalized care by tailoring treatment to the specific needs of each patient.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is one of the most prevalent respiratory disorders, characterized by recurrent pharyngeal collapses during sleep. This disturbance results in fragmented, nonrestorative sleep. Furthermore, intermittent hypoxemia can lead to both acute and chronic elevation of blood pressure and serves as a significant risk factor for all-cause mortality. OSA symptoms include snoring, unrefreshing sleep, fatigue, excessive sleepiness and nocturnal gasping or choking.

OSA is diagnosed using polysomnography (PSG), during which several parameters are measured throughout the night, including airflow, electroencephalography, electromyography, oxygen desaturation and heart rate. Using these measures, OSA severity is quantified by the apnea-hypopnea index (AHI), capturing the number of apneas and hypopneas per hour of sleep.

The standard treatment for OSA is continuous positive airway pressure (CPAP), which opens the upper airway by creating a pneumatic splint. Alternative treatments include mandibular advancement device (MAD) treatment, which (re)opens the upper airway by protruding the mandible, positional therapy to avoid supine position, drug treatments, hypoglossal nerve stimulation treatment and other surgical treatments. While CPAP is characterized by an overall greater efficacy, adherence might be limited. Non-CPAP treatments are characterized by a higher adherence, yet their efficacy is patient dependent.

Respiration-synchronized hypoglossal nerve stimulation (HNS) is an innovative technique in which the hypoglossal nerve is stimulated to protrude the tongue during inspiration. While HNS has demonstrated clinical efficacy, its impact on the underlying pathophysiological mechanisms of OSA remains insufficiently understood. Five pathophysiological parameters are known to be associated with OSA treatment outcome: site of collapse, upper airway collapsibility, ventilatory control instability (loop gain), muscle responsiveness and arousal threshold. These key pathophysiological traits have also been shown to be associated with HNS treatment outcome.

Currently, only the site of collapse is routinely assessed in clinical practice using drug-induced sleep endoscopy (DISE). The remaining traits, particularly collapsibility, usually require complex overnight pressure-drop studies that are not feasible for routine clinical use. Collapsibility is commonly assessed in research using the critical closing pressure (Pcrit), where a higher Pcrit indicates a more collapsible airway.

A recent technique developed by our research group allows for the assessment of the critical closing pressure (Pcrit) during DISE using a modified nasal mask and CPAP device. While the clinical effectiveness of HNS is proven, its specific effect on upper airway collapsibility is unknown.

This study aims to quantify the effect of HNS on upper airway collapsibility by measuring Pcrit during DISE, both with and without active stimulation. This research is vital for understanding the mechanical effects of HNS therapy and may ultimately improve patient selection and the delivery of personalized medicine for OSA.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Treated with HNS-therapy for OSA (AHI ≥15/hour sleep)
* Capable of giving informed consent
* Baseline polysomnography performed at Antwerp University Hospital

Exclusion Criteria:

* Patients did not receive HNS-therapy at the Antwerp University Hospital
* Central apneas accounting for ≥25% of total apneas during baseline polysomnography
* Known medical history of intellectual disability, memory disorders or current psychiatric disorders (psychotic illness, major depression, or acute anxiety attacks as mentioned by the participant).
* Simultaneous use of other treatment modalities to treat OSA (outside of HNS-therapy)
* Esophageal ulceration, tumors, diverticulitis, bleeding varices, sinusitis, epistaxis, recent nasopharyngeal surgery
* Pregnancy or willing to become pregnant
* Excessive alcohol or drug use (> 20 alcohol units/week or any use of hard drugs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
ΔPcrit | One year after HNS implantation, during the 1-year follow-up DISE (= DISE at baseline & DISE with HNS)
  Change in pharyngeal critical closing pressure (ΔPcrit), between baseline Pcrit and Pcrit with HNS. Both Pcrit measurements will be performed on the same day, during the 1-year follow-up DISE.

SECONDARY OUTCOMES:
ΔPcrit in responders and in non-responders | One year after HNS implantation, during the 1-year follow-up DISE (= DISE at baseline & DISE with HNS)
  ΔPcrit in responders and in non-responders. Treatment responders are defined by the Sher15 criteria (AHI decrease of >50% and total AHI<15/h).
∆AHI from baseline to one-year follow-up | From baseline (PSG at baseline, before implantation of hypoglossal nerve stimulator) to one-year follow-up
  ∆AHI from baseline to one-year follow-up to measure treatment response
Δ%area-of-collapse at the level of the palate, tongue base, lateral walls and epiglottis | One year after HNS implantation, during the 1-year follow-up DISE (= DISE at baseline & DISE with HNS)
  Δ%area-of-collapse at the level of the palate, tongue base, lateral walls and epiglottis, between baseline DISE and DISE with HNS

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lou B, Rusk S, Nygate YN, Quintero L, Ishikawa O, Shikowitz M, Greenberg H. Association of hypoglossal nerve stimulator response with machine learning identified negative effort dependence patterns. Sleep Breath. 2023 May;27(2):519-525. doi: 10.1007/s11325-022-02641-y. Epub 2022 May 27. PMID 35622197
- [Background] Sher AE, Schechtman KB, Piccirillo JF. The efficacy of surgical modifications of the upper airway in adults with obstructive sleep apnea syndrome. Sleep. 1996 Feb;19(2):156-77. doi: 10.1093/sleep/19.2.156. PMID 8855039
- [Background] Bamagoos AA, Cistulli PA, Sutherland K, Ngiam J, Burke PGR, Bilston LE, Butler JE, Eckert DJ. Dose-dependent effects of mandibular advancement on upper airway collapsibility and muscle function in obstructive sleep apnea. Sleep. 2019 Jun 11;42(6):zsz049. doi: 10.1093/sleep/zsz049. PMID 30810164
- [Background] Kazemeini E, Van de Perck E, Dieltjens M, Willemen M, Verbraecken J, Op de Beeck S, Vanderveken OM. Critical to Know Pcrit: A Review on Pharyngeal Critical Closing Pressure in Obstructive Sleep Apnea. Front Neurol. 2022 Feb 22;13:775709. doi: 10.3389/fneur.2022.775709. eCollection 2022. PMID 35273554
- [Background] Kazemeini E, Van de Perck E, Dieltjens M, Willemen M, Verbraecken J, Sands SA, Vanderveken OM, Op de Beeck S. Critical closing pressure of the pharyngeal airway during routine drug-induced sleep endoscopy: feasibility and protocol. J Appl Physiol (1985). 2022 Apr 1;132(4):925-937. doi: 10.1152/japplphysiol.00624.2021. Epub 2022 Feb 3. PMID 35112928
- [Background] Smith PL, Wise RA, Gold AR, Schwartz AR, Permutt S. Upper airway pressure-flow relationships in obstructive sleep apnea. J Appl Physiol (1985). 1988 Feb;64(2):789-95. doi: 10.1152/jappl.1988.64.2.789. PMID 3372436
- [Background] Wellman A, Edwards BA, Sands SA, Owens RL, Nemati S, Butler J, Passaglia CL, Jackson AC, Malhotra A, White DP. A simplified method for determining phenotypic traits in patients with obstructive sleep apnea. J Appl Physiol (1985). 2013 Apr;114(7):911-22. doi: 10.1152/japplphysiol.00747.2012. Epub 2013 Jan 24. PMID 23349453
- [Background] Vanderveken OM, Maurer JT, Hohenhorst W, Hamans E, Lin HS, Vroegop AV, Anders C, de Vries N, Van de Heyning PH. Evaluation of drug-induced sleep endoscopy as a patient selection tool for implanted upper airway stimulation for obstructive sleep apnea. J Clin Sleep Med. 2013 May 15;9(5):433-8. doi: 10.5664/jcsm.2658. PMID 23674933
- [Background] Op de Beeck S, Wellman A, Dieltjens M, Strohl KP, Willemen M, Van de Heyning PH, Verbraecken JA, Vanderveken OM, Sands SA; STAR Trial Investigators. Endotypic Mechanisms of Successful Hypoglossal Nerve Stimulation for Obstructive Sleep Apnea. Am J Respir Crit Care Med. 2021 Mar 15;203(6):746-755. doi: 10.1164/rccm.202006-2176OC. PMID 32970962
- [Background] Eckert DJ, White DP, Jordan AS, Malhotra A, Wellman A. Defining phenotypic causes of obstructive sleep apnea. Identification of novel therapeutic targets. Am J Respir Crit Care Med. 2013 Oct 15;188(8):996-1004. doi: 10.1164/rccm.201303-0448OC. PMID 23721582
- [Background] Strollo PJ Jr, Soose RJ, Maurer JT, de Vries N, Cornelius J, Froymovich O, Hanson RD, Padhya TA, Steward DL, Gillespie MB, Woodson BT, Van de Heyning PH, Goetting MG, Vanderveken OM, Feldman N, Knaack L, Strohl KP; STAR Trial Group. Upper-airway stimulation for obstructive sleep apnea. N Engl J Med. 2014 Jan 9;370(2):139-49. doi: 10.1056/NEJMoa1308659. PMID 24401051
- [Background] Vanderveken OM, Beyers J, Op de Beeck S, Dieltjens M, Willemen M, Verbraecken JA, De Backer WA, Van de Heyning PH. Development of a Clinical Pathway and Technical Aspects of Upper Airway Stimulation Therapy for Obstructive Sleep Apnea. Front Neurosci. 2017 Sep 21;11:523. doi: 10.3389/fnins.2017.00523. eCollection 2017. PMID 28983236
- [Background] Sutherland K, Vanderveken OM, Tsuda H, Marklund M, Gagnadoux F, Kushida CA, Cistulli PA. Oral appliance treatment for obstructive sleep apnea: an update. J Clin Sleep Med. 2014 Feb 15;10(2):215-27. doi: 10.5664/jcsm.3460. PMID 24533007
- [Background] Vena D, Op de Beeck S, Mann D, et al. Pharyngeal site of collapse and collapsibility estimated from airflow predict oral appliance treatment efficacy. Sleep Medicine. 2022;100:S264-S265. doi:https://doi.org/10.1016/j.sleep.2022.05.713
- [Background] Sullivan CE, Issa FG, Berthon-Jones M, Eves L. Reversal of obstructive sleep apnoea by continuous positive airway pressure applied through the nares. Lancet. 1981 Apr 18;1(8225):862-5. doi: 10.1016/s0140-6736(81)92140-1. PMID 6112294
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Gottlieb DJ, Punjabi NM. Diagnosis and Management of Obstructive Sleep Apnea: A Review. JAMA. 2020 Apr 14;323(14):1389-1400. doi: 10.1001/jama.2020.3514. PMID 32286648
- [Background] Marshall NS, Wong KK, Cullen SR, Knuiman MW, Grunstein RR. Sleep apnea and 20-year follow-up for all-cause mortality, stroke, and cancer incidence and mortality in the Busselton Health Study cohort. J Clin Sleep Med. 2014 Apr 15;10(4):355-62. doi: 10.5664/jcsm.3600. PMID 24733978
- [Background] Somers VK, White DP, Amin R, Abraham WT, Costa F, Culebras A, Daniels S, Floras JS, Hunt CE, Olson LJ, Pickering TG, Russell R, Woo M, Young T; American Heart Association Council for High Blood Pressure Research Professional Education Committee, Council on Clinical Cardiology; American Heart Association Stroke Council; American Heart Association Council on Cardiovascular Nursing; American College of Cardiology Foundation. Sleep apnea and cardiovascular disease: an American Heart Association/american College Of Cardiology Foundation Scientific Statement from the American Heart Association Council for High Blood Pressure Research Professional Education Committee, Council on Clinical Cardiology, Stroke Council, and Council On Cardiovascular Nursing. In collaboration with the National Heart, Lung, and Blood Institute National Center on Sleep Disorders Research (National Institutes of Health). Circulation. 2008 Sep 2;118(10):1080-111. doi: 10.1161/CIRCULATIONAHA.107.189375. Epub 2008 Aug 25. No abstract available. PMID 18725495
- [Background] Levy P, Kohler M, McNicholas WT, Barbe F, McEvoy RD, Somers VK, Lavie L, Pepin JL. Obstructive sleep apnoea syndrome. Nat Rev Dis Primers. 2015 Jun 25;1:15015. doi: 10.1038/nrdp.2015.15. PMID 27188535

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT07337239/Prot_SAP_000.pdf
  • Informed Consent Form (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT07337239/ICF_001.pdf